CLINICAL TRIAL: NCT01045252
Title: Study of Hemodynamics of Healthy Neonates and Those With Congenital Heart Diseases and Sepsis by Echocardiography and USCOM
Brief Title: Study of Hemodynamics of Neonates by Echocardiography and USCOM
Acronym: HNEU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Shaoru He, Guangdong General Hospital
Other Study IDs: CGGHHSR1132
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Sepsis; Congenital Heart Disease
Keywords: hemodynamics; neonatal
MeSH Terms: conditions — Sepsis; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- congenital heart disease: Neonates that are enrolled in the NICU and are confirmed of congenital heart diseases.
- sepsis: Neonates that are enrolled in the NICU and are diagnosed as sepsis.
- Health: Neonates that are enrolled in the NICU and have no congenital heart diseases and sepsis.

SUMMARY:
The purpose of this study is to evaluate the hemodynamic values of neonates that are healthy and those with various congenital heart diseases and sepsis by using echocardiography and USCOM.

DETAILED DESCRIPTION:
Echocardiography is a diagnostic tool for congenital heart disease.However,it requires skilled specialists to perform it and is a little expensive.Besides,it is too big to move to the bedside easily.USCOM is another newly choice to evaluate hemodynamic values in recent years.This study will compare the hemodynamic values of neonates that are healthy and those with congenital heart diseases and sepsis by using echocardiography and USCOM.

ELIGIBILITY:
Inclusion Criteria:

* neonatal
* congenital heart disease
* sepsis

Exclusion Criteria:

* aged more than thirty days

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients enrolled in the NICU of Guangdong General Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shaoru He, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China